CLINICAL TRIAL: NCT06631521
Title: Neoadjuvant Darolutamide and Relugolix Combination Preceding Radical Prostatectomy for High Risk Localized and Locally Advanced Prostate Cancer: A Phase I/Ib Trial
Brief Title: Neoadjuvant Darolutamide and Relugolix Combination Preceding Radical Prostatectomy for Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Bayer (Industry); Sumitomo Pharma Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR-US-00295; 2077841 (Other: AdventHealth Orlando)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Prostate CA; Prostate Cancer (Adenocarcinoma); Prostate Cancer Surgery
Keywords: Prostate Cancer; High-Risk Prostate Cancer; Neoadjuvant Therapy; Radical Prostatectomy; Darolutamide; Relugolix; Androgen Receptor Antagonists; Gonadotropin-Releasing Hormone Antagonists; Clinical Trial Phase I/Ib; PSA Response
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — darolutamide; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination Therapy Arm (Experimental): This arm is designed to evaluate the safety and feasibility of the combination therapy using darolutamide and relugolix as neoadjuvant treatment before radical prostatectomy (RP) in patients with high-risk prostate cancer (PCa).
  Interventions: Drug: Darolutamide; Drug: Relugolix; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Darolutamide — 600 mg (two 300 mg tablets) taken orally twice daily.
  Other Names: Nubeqa; BAY 1841788
Drug: Relugolix — A loading dose of 360 mg on the first day, followed by 120 mg taken orally once daily.
Procedure: Radical Prostatectomy — Performed at least 48 hours and within 2 weeks after the completion of neoadjuvant therapy.

SUMMARY:
The goal of this clinical trial is to determine the safety and feasibility of a new combination of darolutamide and relugolix as neoadjuvant therapy preceding radical prostatectomy (RP) for high-risk prostate cancer (PCa) in adult males.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate
2. ECOG performance status 0-1
3. Ability to swallow oral medications and comply with study procedures and requirements.
4. Males ≥18 years
5. Participants must have adequate organ and marrow function as below:

   1. Absolute neutrophil count (ANC) ≥1,500/mm3 or ≥1.5 x 109/L;
   2. Platelets ≥100,000/mm3 or ≥100 x 109/L;
   3. Hemoglobin ≥8 g/dL (may have been transfused).
   4. Estimated creatinine clearance ≥30 mL/min as calculated using the Cockcroft-Gault equation.
   5. Total serum bilirubin <1.5 x upper limit of normal (ULN), less than 2.0 x ULN if suspected Gilbert's syndrome;
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN.
6. Must be a candidate for RP
7. Clinical stage cT2-4, N0-1
8. Mandatory to identify tumor availability (≥10 FFPE slides, 5 µM thickness & 1 stained H&E slide OR tumor block)
9. High-risk PCa defined as one of the following-

   * Gleason score (GS) ≥ 4 + 3 with ≥ 6 positive systematic biopsies (SB)
   * GS ≥ 4 + 3 with ≥ 3 SB and prostate-specific antigen (PSA) ≥ 20 ng/mL
   * GS ≥ 9 in ≥ 1 SB or targeted biopsies (TB) -≥ 2 SB or TB with continuous GS ≥ 8, each with ≥ 80% involvement.

Exclusion Criteria:

1. Histologic variants including neuroendocrine differentiation, small cell, sarcomatoid, ductal adenocarcinoma, squamous or transitional cell carcinoma) comprising more than 50% of the sample as determined by pathology review
2. Participants who have had chemotherapy or radiotherapy within 4 weeks prior to planned cycle 1 day 1 of study treatment.
3. Participants who have received anti-neoplastic intervention or experimental antineoplastic therapy within 14 days of planned cycle 1 day 1 of study therapy.
4. Participants who are receiving any other investigational agents.
5. Participants who have previously received darolutamide, relugolix, LHRH agonist/antagonist or another novel androgen blocking therapy (abiraterone, apalutamide, enzalutamide) within 1 year are excluded (prior bicalutamide that was discontinued ≥14 days prior to planned cycle 1 day 1 is allowed).
6. Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e. have residual toxicities ≥Grade 2) with the exception of alopecia.
7. Any of the following within 6 months before planned cycle 1 day 1 of study therapy:

   * Stroke
   * Myocardial infarction
   * Severe/unstable angina pectoris
   * Coronary/peripheral artery bypass graft
   * Congestive heart failure New York Heart Association (NYHA) Class III or IV.
8. Known or suspected contraindications, hypersensitivity or allergy to darolutamide or relugolix or to any of their excipients.
9. Participants with hepatitis C, hepatitis B or human immunodeficiency (HIV) who are on anti-viral therapy that has the potential to interact with darolutamide or relugolix.
10. Participants treated with drugs known to be strong inhibitors and/or inducers of cytochrome P450 3A4 (CYP3A4) and the treatment cannot be discontinued or switched to a different medication at least 5 half-lives prior to starting study drug.
11. NOTE: precaution is warranted with concomitant use of agents with a narrow therapeutic index that are substrates of P-gp, BCRP and OCT1.
12. The participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance less than 30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
13. Concurrent active malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of the investigational regimen. Patients with non-melanomatous skin cancer, superficial bladder cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are permitted to enroll.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing therapy without severe adverse events. | From enrollment, up to 8 weeks after radical prostatectomy.
Number of patients experiencing treatment-related adverse events using CTCAE version 5.0. | From enrollment, up to 8 weeks following radical prostatectomy (RP)

SECONDARY OUTCOMES:
Objective Radiographic Response | From enrollment, up to 12 weeks (end of neoadjuvant therapy).
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes in millimeters (mm). Response refers to the reduction in tumor size according to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) criteria (Complete Response, Partial Response, Stable Disease, or Progressive Disease).
Prostate-specific antigen (PSA) Response | From enrollment, up to 8 weeks after radical prostatectomy.
  The unit of measure is nanograms per milliliter (ng/mL). A PSA response is defined as a decline of ≥50% from baseline levels.
Plasma Concentration of Darolutamide and Relugolix | From enrollment, up to Day 1 of Cycle 3 (Each cycle is 28 days).
  This measure involves assessing the plasma concentration of darolutamide and relugolix at specified time points to determine their pharmacokinetic profiles. Units of measure: Concentration in nanograms per milliliter (ng/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No